## **PROTOCOL TITLE:**

Individualizing Surveillance Mammography for Older Breast Cancer Survivors

## PRINCIPAL INVESTIGATOR:

Rachel A Freedman, MD, MPH
Medical Oncology
617-632-3800
Rachel freedman@dfci.harvard.edu

## **VERSION NUMBER:**

Version 3

NCT03865654

**DATE:** 

07/01/2020



Statistical Analysis Plan:

Pre-visit patient surveys collected demographics, health literacy, numeracy, and preferences for decision-making roles. *Post-visit* surveys included general guide feedback (e.g., length, clarity). Both surveys inquired about intentions for mammography plus past and current (study visit) experiences and comfort level with life expectancy discussions.

From *post-visit* clinician surveys, in addition to acceptability, we described clinician responses for each participating patient for questions that were relevant to a particular patient (e.g., "What did you recommend in terms of mammograms for *this* patient?", "Did you discuss the pros [and cons] of mammography"). In addition to descriptive analyses and extraction of explanatory comments (when provided), we used t-tests to examine changes in patient decisional conflict around mammography from the pre- and post-survey to inform design of a future trial of the guide. All analyses were conducted using SAS.

